CLINICAL TRIAL: NCT07091929
Title: A Randomized, Double-Blind, Placebo-Controlled, Single-Dose Escalation Phase Ib Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Profile, Immunogenicity, and Preliminary Efficacy of SGC001 in Chinese Patients Scheduled to Undergo Percutaneous Coronary Intervention for Anterior ST-segment Elevation Myocardial Infarction
Brief Title: A Research Study to Evaluate the Safety and Preliminary Efficacy of SGC001 in Patients With Myocardial Infarction
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Sungen Biomedical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SG-SGC001-102
Record Dates: First submitted 2025-06-24; First posted 2025-07-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Anterior Myocardial Infarction
MeSH Terms: conditions — Anterior Wall Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SGC001 (Experimental): Enrolled anterior STEMI patients will receive standard clinical treatment and a single dose of SGC001 on Day 1 (D1) according to their randomized dosing group. The study drug should be administered within 6 hours after the onset of acute myocardial infarction symptoms, with earlier administration preferred. The intravenous injection will be administered over 10 minutes.
  Interventions: Drug: SGC001
- Placebo (Placebo Comparator): Enrolled anterior STEMI patients will receive standard clinical treatment and a single dose of placebo on Day 1 (D1) according to their randomized dosing group. The study drug should be administered within 6 hours after the onset of acute myocardial infarction symptoms, with earlier administration preferred. The intravenous injection will be administered over 10 minutes.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SGC001 — The single dose should be administered within 6 hours after the onset of acute myocardial infarction symptoms, with earlier administration preferred. The intravenous injection should be administered over 10 minutes.
  Arms: SGC001
Drug: Placebo — The single dose should be administered within 6 hours after the onset of acute myocardial infarction symptoms, with earlier administration preferred. The intravenous injection should be administered over 10 minutes.
  Arms: Placebo

SUMMARY:
The research study is being done to see if SGC001 can be used to treat people scheduled to undergo percutaneous coronary intervention for Anterior ST-segment Elevation Myocardial Infarction. SGC001 might reduce the infarct size and inhibited inflammation, thereby preventing the incidence of major adverse cardiovascular events(MACE) events. Participants will either get SGC001 (active medicine) or placebo (a dummy medicine which has no effect on the body). Which treatment participants get is decided by chance. The chance of getting SGC001 or placebo is the same. The participant was administered intravenously once. SGC001 is not yet approved in any country or region in the world. It is a new medicine that doctors cannot prescribe.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18~75 years (both inclusive)
2. Anterior STEMI, defined as: (a) Persistent chest pain or discomfort > 30 minutes; AND (b) Persistent ST-segment elevation ≥0.1 mV in ≥2 contiguous precordial leads (V1-V6) on the admission ECG, with ≥0.2 mV required in leads V2 and V3; OR, if （a）clinical symptoms are atypical, (c) a positive point-of-care cardiac troponin test is required.
3. Ability to receive study drug administration within 6 hours of symptom onset, as assessed by the investigator;
4. Subjects who fully understand the purpose, nature, method, and potential adverse reactions of the trial, and who voluntarily sign the informed consent form and agree to participate in the study;

Exclusion Criteria:

1. Individuals with the following medical histories:

   1. Myocardial infarction and coronary revascularization
   2. Cardiopulmonary resuscitation
   3. Stroke within 6 months before the first dose
   4. Aortic dissection
2. Individuals who received thrombolytic therapy;
3. Individuals who have recent febrile infection, requiring systemic treatment;
4. Individuals with cardiogenic shock or hemodynamic instability (such as severe arrhythmia), including systolic blood pressure <90 mmHg;
5. Individuals with clear diagnosis of acute heart failure (Killip grade ≥ III, Killip grade is detailed in appendix);
6. Individuals who cannot undergo cardiovascular magnetic resonance (CMR) testing or are known to be allergic to any radio-contrast agent;
7. Individuals who have participated in other drug clinical studies and received other clinical trial drugs within 1 months prior to receiving the investigational drug;
8. Individuals with the following medical histories:

   1. severe liver and renal insufficiency;
   2. Patients with malignant tumors or previous history of malignant tumors;
   3. Severe autoimmune disease requiring therapeutic intervention;
9. Women of childbearing potential (WOCBP) or men who plan to father a child or whose partners plan to become pregnant from screening until 3 months after receiving the investigational product; pregnant or lactating women;
10. Any other circumstance that, in the judgement of the investigator, may affect the ability of the subject to provide informed consent or to follow the trial protocol, or where the subject's participation in the trial may affect the outcome of the trial or his or her safety.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-07-18 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Adverse events (AE), Serious adverse events (SAE) | From randomisation to end-of-study (up to 30 days)
  Adverse events (AE), Serious adverse events (SAE)
Recommended Phase 2 dose (RP2D) | From randomisation to end-of-study (up to 30 days)
  Determination of the Recommended Phase II Dose

SECONDARY OUTCOMES:
Peak Concentration (Cmax) | From randomisation to end-of-study (up to 30 days)
  Peak Concentration (Cmax)
Time to Maximum Concentration (Tmax) | From randomisation to end-of-study (up to 30 days)
  Time to Maximum Concentration (Tmax)
Area under the plasma concentration-time curve from time zero to the last quantifiable rime point after administration (AUC0-t) | From randomisation to end-of-study (up to 30 days)
  Area under the plasma concentration-time curve from time zero to the last quantifiable rime point after administration (AUC0-t)
Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf) | From randomisation to end-of-study (up to 30 days)
  Area under the plasma concentration-time curve from time zero to infinity (AUC0-inf)
Elimination half-life (t1/2) | From randomisation to end-of-study (up to 30 days)
  Elimination half-life (t1/2)
Elimination rate constant (λz) | From randomisation to end-of-study (up to 30 days)
  Elimination rate constant (λz)
Clearance (CL) | From randomisation to end-of-study (up to 30 days)
  Clearance (CL)
Volume of distribution (Vz) | From randomisation to end-of-study (up to 30 days)
  Volume of distribution (Vz)
Myocardial infarction area percentage[Efficacy endpoints] | From randomisation to end-of-study (up to 30 days)
  Ratio of infarct area to left ventricular area
Absolute myocardial infarction area | From randomisation to end-of-study (up to 30 days)
  Absolute myocardial infarction area
Microvascular occlusion area | From randomisation to end-of-study (up to 30 days)
  Microvascular occlusion area
Left ventricular ejection fraction (LVEF)[Efficacy endpoints] | From randomisation to end-of-study (up to 30 days)
  Left ventricular ejection fraction (LVEF)
Left ventricular end-systolic volume (LVESV)[Efficacy endpoints] | From randomisation to end-of-study (up to 30 days)
  Left ventricular end-systolic volume (LVESV)
Left ventricular end-diastolic volume (LVEDV)[Efficacy endpoints] | From randomisation to end-of-study (up to 30 days)
  Left ventricular end-diastolic volume (LVEDV)
Creatine kinase isoenzyme MB mass (CK-MBmass)[Efficacy endpoints] | From randomisation to end-of-study (up to 30 days)
  Creatine kinase isoenzyme MB mass (CK-MBmass)
High-sensitivity troponin I (hsTnI)[Efficacy endpoints] | From randomisation to end-of-study (up to 30 days)
  High-sensitivity troponin I (hsTnI)
Survival[Efficacy endpoints] | From randomisation to end-of-study (up to 30 days)
  Survival
Qualitative detection of anti-drug antibodies in serum（Anti-drug antibody (ADA)） | From randomisation to end-of-study (up to 30 days)
  Qualitative detection of anti-drug antibodies in serum by ELISA, followed by calculation of the positivity rate as the number of positive samples divided by the total number of samples

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, Bachelor, Study Director — The Second Affiliated Hospital of Harbin Medical University
Locations (4):
- China (4):
  - Beijing Anzhen Hospital Capital Medical University, Beijing, Beijing Municipality
  - The 2nd Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Linfen Central Hospital, Linfen, Shanxi
  - Teda International Cardiovascular Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will be shared when necessary